CLINICAL TRIAL: NCT03331250
Title: A Pilot Phase 2 Study of Eribulin in Angiosarcoma and Epithelioid Hemangioendothelioma (EHE)
Brief Title: Eribulin in Angiosarcoma and Epithelioid Hemangioendothelioma (EHE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Gregory Cote, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-355
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Angiosarcoma; Epithelioid Hemangioendothelioma
Keywords: Epithelioid hemangioendothelioma (EHE); Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma; Hemangioendothelioma, Epithelioid | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eribulin (Experimental): * Eribulin administered twice per cycle intravenously
  * Each cycle contains 21 days
  * Dosing is per the FDA label for other cancers
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — It may work by preventing the cancer cells from dividing and eventually cause the tumor cells to die
  Other Names: Halaven

SUMMARY:
This research study is studying a drug as a possible treatment for Angiosarcoma or Epithelioid hemangioendothelioma (EHE).

-The drug involved in this study is Eribulin

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Eribulin for your specific disease but it has been approved for other uses.

In this research study, the investigators are studying how safe and effective eribulin is in participants with Angiosarcoma or EHE.

Eribulin was created to mimic the structure of a chemical that is released from a sea sponge. The investigators believe that this drug has anti-cancer effects on tumors by blocking proteins called microtubules, among other functions. It may work by preventing the cancer cells from dividing and eventually cause the tumor cells to die similar to other drugs that target microtubules

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced angiosarcoma, treated with at least one prior systemic therapy where no standard of care curable therapy is available OR metastatic or locally advanced malignant and progressive epithelioid hemangioendothelioma (EHE).
* A maximum of 5 EHE patients will be accrued on this study
* Archival tissue confirming the diagnosis must be reviewed by BWH/DFCI/MGH pathology.
* Progression on at least one prior systemic therapy or progression during an observation phase of no anti-cancer therapy within the prior 3 months; prior taxanes are allowed
* Participants must have measurable disease by RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Age > 18 years.
* ECOG performance status ≤2
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Baseline QTcF < grade 2
* The effects of Eribulin on the developing human fetus are unknown. For this reason and because of the risk of teratogenicity, women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation, and 4 months after completion of Eribulin administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Eribulin administration.
* Willingness to undergo serial tumor biopsies before and on treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C), immunotherapy within 3 weeks, targeted therapies (e.g. small molecule inhibitors such as pazopanib) within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Not clinically significant or clinically stable adverse events from prior therapy (e.g. immunotherapy related hypothyroidism or insulin-dependent diabetes stable on medication or TKI-related hypertension or rash etc.) is allowed.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases and/or leptomeningeal disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to eribulin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NYHA Class II), unstable angina pectoris or myocardial infarction within 6 months of enrolment, serious or life-threatening cardiac arrhythmia, subjects with a high probability of Long QT syndrome or QTcF prolongation of > 501 mcsec (grade 2) on at least two separate ECG following correction of any electrolyte imbalance or psychiatric illness/social situations that would limit compliance with study requirements.
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Eribulin. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2026-02-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cote, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Eribulin: * Eribulin administered twice per cycle intravenously
  * Each cycle contains 21 days
  * Dosing is per the FDA label for other cancers
  Eribulin: It may work by preventing the cancer cells from dividing and eventually cause the tumor cells to die
Period: Overall Study
Arm/Group | Eribulin
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eribulin
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 61.7 [42.3 to 76.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as the percentage of patients who achieved a partial response or complete response by RECIST 1.1. Tumor imaging studies were completed using either CT (Computed Tomography) or MRI (Magnetic resonance imaging). The modality chosen for any individual patient was the same from baseline until the end of their time on study.
  Per RECIST v 1.1, complete response (CR) is defined as the disappearance of all target lesions and the reduction in any pathological lymph nodes in short axis to less than 10 mm. Partial response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions compared with baseline. Progressive disease (PD) is defined as a 20% increase (5+ mm absolute increase) compared with the smallest sum on study. Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor PD.
Time Frame: 2 years
Population: One patient out of the 13 who enrolled withdrew from the study before completing any cycles of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin
Number analyzed (Participants) | 12
Participants | 4

2. Secondary Outcome: Progression Free Survival
Time Frame: 4 years
Reporting Status: Not Posted

3. Secondary Outcome: Disease Control Rate
Description: Objective Response plus Stable Disease Rate at 24 weeks
Time Frame: 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Treatment Related Adverse Events
Description: Summary of the treatment related adverse events experienced by study participants as assessed by Common Terminology Criteria for Adverse Events (CTCAE v4)
Time Frame: 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All AEs were collected from cycle 1 day 1 until either 28 days after the subject's last dose (an average 37 weeks), or resolution/stabilization of an AE if continuing beyond 28 days.
Arm/Group | Eribulin
All-Cause Mortality (participants affected / at risk) | 11/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin (N=13)
Anemia (Blood and lymphatic system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Periorbital infection (Infections and infestations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin (N=13)
Abdominal pain (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 2
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Burn (Injury, poisoning and procedural complications) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 4
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Neutrophil count decreased (Investigations) | 3
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Periorbital infection (Infections and infestations) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6
Presyncope (Nervous system disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin infection (Infections and infestations) | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Watering eyes (Eye disorders) | 2
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03331250/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT03331250/ICF_001.pdf